CLINICAL TRIAL: NCT00265928
Title: VELCADE (Bortezomib) for Injection - Phase II Study of Bortezomib and Rituximab in Relapsed or Refractory Non-Hodgkin's Lymphoma
Brief Title: Bortezomib and Rituximab in Treating Patients With Relapsed or Refractory B-Cell Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawn for poor accrual
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000459747; UVACC-HIC-12077; UVACC-PRC-36805; MILLENNIUM-X05181; MILLENNIUM-LYMPHOMA2
Record Dates: First submitted 2005-12-14; First posted 2005-12-15 (Estimated); Last update posted 2008-01-28 (Estimated); Status verified 2007-01

CONDITIONS: Lymphoma
Keywords: extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; splenic marginal zone lymphoma; recurrent adult diffuse small cleaved cell lymphoma; nodal marginal zone B-cell lymphoma; Waldenstrom's macroglobulinemia
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Waldenstrom Macroglobulinemia | interventions — Bortezomib; Rituximab; Immunization, Passive; Biological Therapy; Antibodies, Monoclonal

INTERVENTIONS:
Drug: bortezomib
Drug: rituximab
Procedure: antibody therapy
Procedure: biological therapy
Procedure: enzyme inhibitor therapy
Procedure: monoclonal antibody therapy

SUMMARY:
RATIONALE: Bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Giving bortezomib together with rituximab may be an effective treatment for non-Hodgkin's lymphoma.

PURPOSE: This phase II trial is studying how well giving bortezomib together with rituximab works in treating patients with relapsed or refractory B-cell non-Hodgkin's lymphoma, including Waldenstrom's macroglobulinemia.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the safety and tolerability of bortezomib and rituximab in patients with relapsed or refractory, B-cell non-Hodgkin's lymphoma.
* Determine the overall response rate (partial response, complete response unconfirmed, and complete response) in these patients.

Secondary

* Estimate the duration of response in patients treated with this regimen.
* Estimate the time to disease progression in patients treated with this regimen.

OUTLINE: This is an open-label study.

Patients receive bortezomib IV over 3-5 seconds once weekly in weeks 1-4 and rituximab IV over 5-6 hours once weekly in weeks 1-5*. Treatment repeats every 5 weeks for 2 courses. Patients achieving stable disease or better receive an additional 4 courses of bortezomib alone.

NOTE: *Patients receive rituximab in weeks 1-3 only during course 2 of treatment.

After completion of study treatment, patients are followed periodically for at least 18 months.

PROJECTED ACCRUAL: A total of 46 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed B-cell non-Hodgkin's lymphoma (NHL) including the following subtypes:

  * B-cell small lymphocytic lymphoma
  * Marginal zone lymphoma (extranodal, nodal, or splenic)
  * Grade 1-3 follicular lymphoma
  * Mantle cell lymphoma
  * Waldenstrom's macroglobulinemia
* Bidimensionally measurable disease by CT scan with ≥ 1 lesion measuring > 1.5 cm in a single dimension
* Relapsed or refractory disease after prior antineoplastic therapy, meeting 1 of the following criteria:

  * No response to prior treatment
  * Relapsed disease after prior therapy
* Confirmed CD20-positive disease by immunohistochemistry on biopsy specimen

  * Prior transformation allowed provided there is no evidence of aggressive histology on recent biopsy
* No chronic lymphocytic lymphoma with absolute lymphocyte count > 5,000/mm³
* No CNS involvement

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm^3 (≥ 1,000/mm³ if due to extensive bone marrow involvement with NHL or splenomegaly)
* Absolute lymphocyte count ≤ 5,000/mm³ (except mantle cell lymphoma with a leukemic phase)
* Platelet count ≥ 50,000/mm^3
* Bilirubin ≤ 2.0 mg/dL
* AST and ALT ≤ 2.5 times upper limit of normal (ULN) (4 times ULN if liver involvement with NHL)
* Creatinine ≤ 2.0 mg/dL
* Not pregnant or nursing
* Negative pregnancy test
* Fertile male and female patients must use effective contraception during study
* No serious nonmalignant disease
* No active infection
* No peripheral neuropathy ≥ grade 2 within past 14 days
* No myocardial infarction within the past 6 months
* No New York Heart Association class III or IV heart failure
* No uncontrolled angina pectoris
* No severe uncontrolled ventricular arrhythmias
* No EKG evidence of acute ischemia or active conduction system abnormalities
* Any EKG abnormality must be documented as not medically relevant
* No hypersensitivity to bortezomib, boron, or mannitol
* No known anaphylaxis or immunoglobulin E-mediated hypersensitivity to murine proteins or any component of rituximab (including polysorbate 80 and sodium citrate dehydrate)
* No known infection or exposure to HIV
* No serious psychiatric or medical illness that would preclude study participation
* No active hepatitis B infection
* No other primary malignancy requiring active treatment
* More than 4 weeks since prior significant traumatic injury

PRIOR CONCURRENT THERAPY:

* At least 3 weeks since prior and no concurrent radiotherapy
* More than 4 weeks since prior major surgery or open biopsy

  * Other diagnostic surgery allowed
* More than 4 weeks since prior cytotoxic chemotherapy (6 weeks for nitrosoureas)
* At least 3 months since prior unconjugated monoclonal antibody therapy
* At least 10 weeks since prior radioimmunoconjugates or toxin immunoconjugates (e.g., iodine I 131 tositumomab [Bexxar] or ibritumomab tiuxetan [Zevalin])
* More than 2 weeks since prior investigational agent
* No prior bortezomib
* No concurrent systemic corticosteroid at greater than the equivalent dose of 20 mg/day of prednisone, unless for treatment of allergic reactions to CT scan dye
* No concurrent major surgery
* No other immunosuppressive agents, unless for treatment of allergic reactions to CT scan dye
* No other concurrent antilymphoma agents
* No other concurrent investigational agent

  * Concurrent participation in another nontreatment study allowed if it does not interfere with participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: John Densmore, MD, Study Chair — University of Virginia
Locations (1):
- University of Virginia Cancer Center at UV Health System, Charlottesville, Virginia, United States